CLINICAL TRIAL: NCT05974774
Title: Intermittent Androgen Deprivation Therapy in the Era of AR Pathway Inhibitors; a Phase 3 Pragmatic Randomized Trial.
Brief Title: Intermittent Androgen Deprivation Therapy in the Era of AR Pathway Inhibitors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Cancer Trials Ireland (Network); UNICANCER (Other); Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 2238
Record Dates: First submitted 2023-06-26; First posted 2023-08-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Metastatic hormone-naïve prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 7-iodo-8-hydroxy-3-methyl-1-(4-azidophenyl)-2,3,4,5-tetrahydro-1H-3-benzazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - continuous treatment (Active Comparator): Arm A (cMAB): ADT (LHRH agonist or antagonist) + ARPI (abiraterone or enzalutamide or apalutamide or darolutamide) continuously until start of a new anti-cancer therapy.
  Interventions: Drug: cMAB
- Arm B - intermittent treatment (Experimental): Arm B (iMAB): no further treatment, including ADT and ARPI; decision to restart ADT (LHRH agonist or antagonist) and the initial ARPI (abiraterone, enzalutamide, apalutamide or darolutamide) is left at Investigator discretion.
  Interventions: Drug: iMAB

INTERVENTIONS:
Drug: iMAB — no treatment until significant PSA increase as per treating physician at which point patient restarts ADT (LHRH agonist or antagonist) + ARPI (abiraterone or enzalutamide or apalutamide or darolutamide). Once PSA < 0.2 ng/mL, treatment stops again.
  Other Names: intermittent maximum androgen blockade
  Arms: Arm B - intermittent treatment
Drug: cMAB — LHRH agonist or antagonist + ARPI (abiraterone or enzalutamide or apalutamide or darolutamide)
  Other Names: continuous maximum androgen blockade
  Arms: Arm A - continuous treatment

SUMMARY:
This study addresses the global topic of treatment optimization, i.e. achieving similar benefit while reducing the duration of treatment, hence hoping to decrease the burden of side-effects, improve quality-of life and reduce resource utilization.

The primary goal of de-escalation is to investigate whether using an intermittent regime results in a similar OS to continuous treatment.

DETAILED DESCRIPTION:
Prostate cancer is known to be dependent on testicular and adrenal androgens and the earliest identified treatments were the suppression of the body's production of testosterone. Then came the development of drugs able to block the androgen receptors that multiplied on the cancer cell membranes. The combination of these drugs presently approved by the EMA for first line treatment of mHNPC are understood to be given maximum androgen blockage and to be used until progression. All have been shown to positively impact overall survival. For patients, however, the consequences of continuous intensified MAB, and thereby testosterone suppression, have impacted their quality of life, especially in the form of fatigue, emotional distress, decrease of libido and loss of sexual function. This is in addition to toxicities linked to the mechanisms of these drugs which include cardiovascular diseases, cognitive effects and loss of bone mineral density.

Treatment optimization is rarely addressed by clinical trials run for registration purposes. Toxicity is subsumed under efficacy and keeping the cancer at bay or controlled at any cost. Overall patient experience is not taken into account when determining what is an acceptable trade-off. Intermittent treatment or drug holiday are options to manage drug toxicities but longer off-treatment periods remain rare due to the fear of losing efficacy.

Prostate cancer is an ideal setting to study the benefits of intermittent treatment as PSA levels have been shown to be a good indicator of cancer status. By holding androgen blockade after good PSA response, patients get the opportunity of seeing an improvement in their quality of life as testosterone levels slowly recover. The longer a patient stays off treatment, the more improvements to his overall wellbeing can be felt. Monitoring PSA levels provides an early signal to cancer regrowth and allows for the restart of MAB when it becomes necessary.

While improving the patient's quality of life, there is as yet no indication as to the possible impact of this approach on overall survival. Alternating off/on treatment could delay both the start of the next line of treatment and the development of castration resistance but the absence of constant androgen suppression could also have the opposite effect and precipitate new alternatives to cancer cells testosterone dependence.

This trial will randomize patients to either continue with their treatment as prescribed or to stop treatment until PSA levels indicate the necessity of restarting suppression. The latter group can stop treatment again when PSA levels reaches 0.2 ng/mL or lower. There is a need to investigate whether the benefit to patient's lives of holding long-term treatment will outweigh the risks of shortening overall survival. This trial is being done to allow both patients and their treating teams to have the data needed to make an informed decision on the best treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with ADT and an ARPI for mHNPC for 6-12 months and presenting with a PSA ≤ 0.2 ng/mL Note: Patient may have received docetaxel and radiotherapy of the prostate and metastases Note: Patients with synchronous or metachronous metastases, high volume/risk or low volume/risk who fulfil the criteria can be included.
* Before patient 's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Patients with M1a on modern imaging technique (PET-Choline or -PSMA or Whole Body MRI) for whom radiation therapy and 2-3 years of hormone therapy is planned
* Patients who underwent or will undergo a bilateral orchiectomy
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment for this trial
* Patients who have received a systemic anti-prostate cancer treatment not approved by EMA together with MAB or a radical prostatectomy for M1 disease
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2035-05-23 (Estimated); Study Completion 2039-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 10 years from randomisation
  the overall survival (OS) using an iMAB regimen is non-inferior to continuous treatment.
proportion of patients who do not restart their hormonal therapy within 1 year of interrupting their MAB therapy (given as part of the induction phase) | 1 year from stopping the MAB therapy
  proportion of patients who do not restart within 1 year of interrupting their MAB therapy (given as part of the induction phase) is not less than 70%

SECONDARY OUTCOMES:
occurrence of adverse events | 10 years from randomisation
  Safety according to the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for toxicity and Serious Adverse Event reporting.
Time spent on MAB treatment | 10 years from randomisation
  the overall time in months that the patient was on MAB treatment
Time to next systemic prostate cancer therapy | 10 years from randomisation
  the overall time in months until the patient began the next systemic prostate cancer therapy
The magnitude of change in HRQoL | 60 months from randomisation
  The magnitude of change in HRQoL in terms of physical functioning from EORTC QLQ-C30
The magnitude of change in HRQoL | 60 months from randomisation
  The magnitude of change in HRQoL in terms of sexual activity, physical fatigue and pain characteristics from the IL249 item list; To cover all important HRQoL domains and to have more granularity on some of the selected domains, additional HRQoL concepts are searched in the EORTC item library. This resulted in the inclusion of an additional scale that measures the pain characteristics.
  The selected scale and corresponding items address the pain characteristics (the nature of the pain: constant versus intermittent and whether the pain can be relieved by pain medications)
health utility derived from the QLQ-C30 questionnaires data | 10 years from randomisation
  Health utility derived from patient reported QLQ-C30 data and patient demographics;Health utilities summarize a patient's overall health status, and this parameter can be applied in cost-effectiveness analyses. Published mapping algorithms can be used to calculate health utility based on the collected QLQ-C30 data, either directly or indirectly. The indirect algorithms first maps QLQ-C30 scores to European Quality-of-Life-5 Dimensions (EQ-5D) scores and then to health utility scores. The collected HRQoL data using QLQ-C30 will be mapped first to EQ-5D scores using an established mapping approach from the literature, and then further translated to health utility values for each study subject and at each assessment of HRQoL, taking into account published national value sets for this conversion.
Prostate cancer specific survival | 10 years from randomisation
  Prostate cancer specific survival will be computed from the date of randomization to the date of death due to prostate cancer. Participants who died from other causes will be considered as having a competing event at this time. Participants who are still alive at the analysis cut-off date are censored at the last date known to be on protocol treatment (before the cut-off date).

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Tombal, Prof, Study Chair — Cliniques Universitaires de Saint Luc; Silke Gillessen, Prof, Study Chair — Oncology Institute of Southern Switzerland - Ospedale San Giovanni
Locations (9):
- University Hospitals Copenhagen - Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Centre Francois Baclesse, Caen
  - Institut Daniel Hollard, Grenoble
  - Clinique La Croix Du Sud, Quint-Fonsegrives
  - CHU de Toulouse - Institut Claudius Regaud - IUCT oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Spain (3):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda